CLINICAL TRIAL: NCT06426940
Title: Prospective Analysis of Anesthesia-Related Peroperative Critical Events in a Tertiary Care Hospital
Brief Title: Anesthesia-Related Peroperative Critical Events
Status: Completed | Type: Observational
Sponsor: Gamze Küçükosman (Other)
Responsible Party: Sponsor-Investigator, Gamze Küçükosman, associate professor, Zonguldak Bulent Ecevit University
Organization: Zonguldak Bulent Ecevit University (Other)
Other Study IDs: SBÜTrabzon
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-05

CONDITIONS: The Frequency of Anesthesia-related Critical Events; Anesthesia-related Intraoperative Critical Events; Anesthesia-related Postoperative Critical Events

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- intraoperative anesthesia-related critical events
  Interventions: Other: anesthesia-related critical events
- postoperative 1 hour (h)anesthesia-related critical events
  Interventions: Other: anesthesia-related critical events

INTERVENTIONS:
Other: anesthesia-related critical events — anesthesia-related critical events

SUMMARY:
Peroperative anesthesia-related critical events (CE) lead to adverse health outcomes in patients. To minimize recurrence of these outcomes, identifying problems causing CEs and obtaining information about their frequency and severity are important. This study aims to determine the frequency of anesthesia-related CEs occurring within intraoperative and postoperative 1 hour (h) in surgical patients at our tertiary care hospital, by system.

ELIGIBILITY:
Inclusion Criteria:

* All patients

Exclusion Criteria:

* intubated outside the operating room
* taken into operation from the intensive care unit (ICU).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Age, gender, ASA (the American Society of Anesthesiologists) risk, surgical clinic, anesthesia method (general/regional/local/sedation/local+sedation), anesthesia and surgery duration of the patients, and anesthesia-related CEs occurring within intraoperative and postoperative 1 h were recorded.
Sampling Method: Non-Probability Sample
Enrollment: 1904 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Prospective Analysis of Anesthesia-Related Peroperative Critical Events in a Tertiary Care Hospital | anesthesia-related intraoperative and within postoperative 1 hour critical events
  This study aims to determine the frequency of anesthesia-related CEs occurring within intraoperative and postoperative 1 hour (h) in surgical patients at our tertiary care hospital, by system.

CONTACTS AND LOCATIONS:
Overall Officials: gamze küçükosman, Principal Investigator — Zonguldak Bulent Ecevit University
Locations (1):
- Gamze Küçükosman, Zonguldak, Zonguldak Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided